CLINICAL TRIAL: NCT04463459
Title: Effect of Vitamin C and Vitamin E in Breast Cancer Patients Undergoing Chemotherapy
Brief Title: Effect of Vitamin C and E in Breast Cancer Patients Undergoing Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Fatisha Khanam, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSMMU/2019/8874
Record Dates: First submitted 2020-06-25; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Vitamin C; Vitamin E; Breast cancer; Chemotherapy; MDA; RBC Glutathione
MeSH Terms: conditions — Breast Neoplasms | interventions — Ascorbic Acid; Vitamin E

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy + Placebo (No Intervention): Patients receiving chemotherapy This group will be received chemotherapy and placebo
- Chemotherapy + Vitamin C + Vitamin E (Active Comparator): Patients receiving vitamin C and E with Chemotherapy This group will be received vitamin C (500 mg) twice daily and vitamin E (400 mg) once daily with chemotherapy for 6 weeks
  Interventions: Drug: Vitamin C, Vitamin E

INTERVENTIONS:
Drug: Vitamin C, Vitamin E — Vitamin C (500mg) twice daily and Vitamin E (400mg) once daily
  Arms: Chemotherapy + Vitamin C + Vitamin E

SUMMARY:
Title:

Effect of Vitamin C and Vitamin E in Breast Cancer patients undergoing Chemotherapy.

Purpose of the study:

The present study has been designed to assess the effects of vitamin C and vitamin E superimposed upon chemotherapeutic agents where the antioxidant vitamin C and vitamin E would be concurrently applied to breast cancer patients.

Method:

The study would be a quasi-experimental study involving breast cancer patients and would be conducted in the Department of Pharmacology and Department of Oncology, BSMMU, from March 2019 to August 2020. A total of 80 breast cancer patients would be selected by abiding selective inclusion and exclusion criteria. After completing necessary formalities including informed written consent of the patients, patient's requisite data will be collected. The diagnosed patients would be randomly allocated into two groups: group A (control group) and group B (intervention group). Group A would consist of 40 patients who will receive chemotherapy and group B would consist of 40 patients who will receive vitamin C (1000 mg) and vitamin E (400 mg) orally daily along with chemotherapy. Both groups would receive treatment for 8 weeks. Comparison between the two groups would be performed through biochemical parameters such as total antioxidant capacity (TAC) and total oxidant status (TOS) at baseline (before vitamin C and vitamin E supplementation) and 6 weeks after intervention by vitamin C and E supplementationtation.

Ethical consideration:

The study will follow the principles of the Declaration of Helsinki and the World Medical Assembly. Patients will be informed about the study in easy language and then informed consent will be taken. This study has no potential risk to the patients. Confidentiality will be strictly maintained.

DETAILED DESCRIPTION:
Breast cancer is a devastating cancer having multifactorial origin. It is the most common cancer and second leading cause of death in women. Every year more than one million breast cancer patients are diagnosed throughout the world and it has been assumed that among them more than 410000 would die due to the disease. In our country due to the absence of official registry records, not much information about breast cancer. 12764 new cases of breast cancer were diagnosed and 6846 women died in Bangladesh in the year 2018. In low- and middle-income countries including Bangladesh due to lower resource settings women with breast cancer may receive inadequate treatment, palliative care or pain relief. The study would be a quasi-experimental study involving breast cancer patients and would be conducted in the Department of Pharmacology and Department of Oncology, BSMMU, from March 2019 to August 2020. A total of 80 breast cancer patients would be selected by abiding selective inclusion and exclusion criteria. After completing necessary formalities including informed written consent of the patients, patient's requisite data will be collected. The diagnosed patients would be randomly allocated into two groups: group A (control group) and group B (intervention group). Group A would consist of 40 patients who will receive chemotherapy and group B would consist of 40 patients who will receive vitamin C (1000 mg) and vitamin E (400 mg) orally daily along with chemotherapy. Both groups would receive treatment for 8 weeks. Comparison between the two groups would be performed through biochemical parameters such as total antioxidant capacity (TAC) and total oxidant status (TOS) at baseline (before vitamin C and vitamin E supplementation) and 6 weeks after intervention by vitamin C and E supplementationtation. Statistical analysis will be obtained by SPSS (Statistical Package for Social Science) version 20. Results will be presented in tables and figures as applicable. Calculated 'P' value may suggest the level of significance (significant at P˂0.05, 0.01 and 0.001). Patients will be informed about the study in easy language and then informed consent will be taken. This study has no potential risk to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patient before starting chemotherapy and will agree to take protocol based chemotherapy.
* Age: 30-70 years.
* Gender: Female.

Exclusion Criteria:

* Patients receiving chemotherapy prior to attend the Department of Oncology, BSMMU.
* Users of any antioxidant nutrient (e g. vitamin A, vitamin C or vitamin E) which can interfere with concentration of endogenous antioxidant estimation.
* Patients with impaired renal and hepatic function.
* Patients with systemic illness such as diabetes, hypertension.
* Presence of any malignancy other than breast cancer.
* Mentally sick patient.
* Smoker.
* Patient suffering from alcohol or substance abuse or dependence.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
To measure the serum level of MDA and RBC glutathione in breast cancer patients receiving chemotherapy and following administration of vitamin C and vitamin E concurrent to chemotherapy. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fatisha Khanam, MBBS, Principal Investigator — BSMMU(Recruting), Dhaka-1000, Bangladesh
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No